CLINICAL TRIAL: NCT04094428
Title: Burden, Mortality and Supply Costs in Intensive Care Unit Patients. Health Services Research.
Brief Title: Burden, Mortality and Supply Costs in Intensive Care Unit Patients
Acronym: PLV_Ulm
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Manfred Weiss, Professor, MD, University of Ulm
Other Study IDs: Anae_ICU_Ulm_PLV
Record Dates: First submitted 2019-09-12; First posted 2019-09-19 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Burden, Dependency; Mortality; End-of-life Care; Intensive Care Unit; Critically Ill Patient; Frailty; Multiple Organ Failure
Keywords: burden; mortality; end-of-life care; intensive care unit; critically ill patient; frailty; Multiple Organ Failure
MeSH Terms: conditions — Frailty; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intensive care unit patient: All intensive care unit patients staying for at least 72 hours on the ICU and patients dying within 72 hours

SUMMARY:
This study systematically observes in a pragmatic trail under real world conditions the association between strategies of therapy (maximal therapy, withhold, withdraw) and treatment success in three endpoint related initial risk groups (high, intermediate, low risk) regarding three endpoints (burden, mortality and supply costs).

DETAILED DESCRIPTION:
This study systematically observes in a pragmatic trail under real world conditions the association between strategies of therapy (maximal therapy, withhold, withdraw) and treatment success in three endpoint related initial risk groups (high, intermediate, low risk) regarding three endpoints (burden, mortality and supply costs).

The 3 endpoints and 3 respective risk groups (high, intermediate, low) are

1. Endpoint burden of care due to Clinical Frailty Scale (Frailty) high 7 - 9 intermediate 5 - 6 low 1 - 4
2. Endpoint mortality due to severity of disease regarding Simplified Acute Physiology Score (SAPS) II score values high SAPS II > 70, suspected mortality > 40% intermediate SAPS II > 40 - 70, suspected mortality 10 - 40% low SAPS II ≤ 40, suspected mortality < 10%
3. Endpoint supply costs due to number of organ systems to be supported or replaced high ≥ 3 organ systems replaced intermediate 1 - 2 organ systems replaced low 0 - 2 organ systems replaced

ELIGIBILITY:
Inclusion Criteria:

* All patients dying on the ICU and all patients staying for at least 72 hours on the ICU

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients admitted to the intensive care unit, mainly surgical and polytraumatized patients
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Burden of care | 18 months
  Organ dysfunctions supported or replaced in numbers
Mortality | 18 months
  Dying patients in numbers
Supply costs | 18 months
  Costs in sum of Simplified Acute Physiology Score (SAPS) II score points over ICU stay; Costs in sum of points of organ support over ICU stay; Costs in Euro reimbursed for the ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Weiss, MD, MBA, Principal Investigator — University Hospital Medical School
Locations (1):
- Department of Anaesthesiology, University Hospital Ulm, Ulm, Germany

IPD SHARING:
Plan to Share IPD: No